CLINICAL TRIAL: NCT00155974
Title: Rapid Vaccination of Hard-to-Reach Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The New York Academy of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 091603; DA017004
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Influenza
Keywords: Influenza; Vaccination; Hard-to-Reach Populations; Urban; Disadvantaged
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Community-based vaccine outreach intervention

SUMMARY:
The purpose of this study is to develop and determine the effectiveness of a multi-level community participatory intervention designed to rapidly immunize hard-to-reach populations, including substance users, within disadvantaged minority communities.

Specific Aims of the project are as follows:

1. To identify the relative contributions of personal factors and structural barriers to immunization status in hard-to-reach populations.
2. To estimate the size of the hard-to-reach population in specified disadvantaged urban communities using venue-based sampling, probability-based sampling, capture-recapture methods and modified Delphi techniques.
3. To compare vaccination rates in hard-to-reach populations between neighborhoods that receive a community-based vaccine outreach intervention versus neighborhoods where vaccines are offered through standard public health programs, using an incremental crossover multilevel community intervention design.

DETAILED DESCRIPTION:
This study follows a quasi-experimental design involving a multilevel community participatory intervention that is designed to rapidly immunize hard-to-reach (HTR) populations in disadvantaged minority communities. Low vaccination coverage among minorities and persons living in and near poverty is a persistent problem that is particularly acute among HTR populations (e.g. injection drug users, elderly shut-ins). Immunization rates are affected by multiple factors including demographics, attitudes about vaccination, health norms, barriers to access, and immunization delivery methods. Efforts to successfully vaccinate HTR populations must address these factors. A community-based program with rapid vaccination can serve as an initial model for emergency preparedness vaccination plans and for future efforts to widely introduce HIV vaccination in disadvantaged urban communities. This project will be conducted by a community-public health partnership in eight disadvantaged neighborhoods within Harlem and the South Bronx in three phases. In Phase 1 we will implement a brief survey assessment of residents in designated neighborhoods to identify current key barriers to immunization faced by the target HTR populations in these neighborhoods. Also, using several estimation methods, we will determine the size of the target populations in the study neighborhoods to establish vaccine needed and to estimate denominators for vaccination rates. In Phase 2, we will implement two waves of a multilevel community intervention trial (developed with input from the survey and community partners). In the first wave, four randomly selected neighborhoods will receive the intervention (i.e., community education, community-organization engagement, and door-to-door influenza vaccination program for eligible groups etc). In the four control communities, target populations will be invited to come for vaccination at specified locations as part of usual public health efforts. In the second vaccination wave, using a crossover design, after updating and revising the approach based on experience from Wave 1, we will implement the intervention in the four control communities; this vaccination wave will be conducted over one week to test the feasibility of rapid vaccination of these populations. Phase 3 of this project will identify the promising elements of the program and develop materials to allow generalizability to other urban areas and to other vaccines (e.g., HIV, HBV, etc).

ELIGIBILITY:
Inclusion Criteria:

The possible participant pool for this project is the adult population (over the age of 18) of 8 circumscribed neighborhoods in East Harlem and South Bronx in NYC. These neighborhoods have a total population of approximately 24,000 people (based on the 2000 US Census) and we anticipate that up to 4,000 may be among the eligible hard-to-reach populations that are the target of this proposal. We will identify eligible populations through a brief survey instrument. During the intervention phase of this study, persons who are eligible to receive influenza vaccination will be offered influenza vaccination. Eligibility criteria for influenza vaccination are the eligibility criteria established by the Advisory Committee on Immunization Practices guidelines. These will be determined as part of the standard data collection instrument. Eligible persons include persons over the age of 65 and persons concurrent comorbidity including immunosuppression (HIV or active injection drug use), chronic pulmonary or cardiovascular disorder (including asthma), or chronic metabolic diseases (including diabetes mellitus, renal or hepatic dysfunction).

Exclusion Criteria:

Exclusion criteria include an allergy to vaccines, an allergy to eggs, inability to provide consent, currently under care of a physician and a plan to receive influenza vaccine in the near-future, or having already received the influenza vaccine during this year (CDC 1999).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000
Dates: Start 2004-02; Study Completion 2005-10

PRIMARY OUTCOMES:
Compare vaccination rates in selected neighborhoods before and after a multilevel community-based participatory intervention trial.

SECONDARY OUTCOMES:
Determine and identify the relative contributions of personal factors and structural barriers to immunization status in hard-to-reach populations.
Estimate the size of the hard-to-reach populations.

CONTACTS AND LOCATIONS:
Overall Officials: David Vlahov, PhD, Principal Investigator — Center for Urban Epidemiologic Studies, The New York Academy of Medicine; Sandro Galea, MD, DrPH, Principal Investigator — Center for Urban Epidemiologic Studies, The New York Academy of Medicine
Locations (1):
- Center for Urban Epidemiologic Studies, The New York Academy of Medicine, New York, New York, United States

REFERENCES:
- [Background] Galea S, Sisco S, Vlahov D. Reducing disparities in vaccination rates between different racial/ethnic and socioeconomic groups: the potential of community-based multilevel interventions. J Ambul Care Manage. 2005 Jan-Mar;28(1):49-59. doi: 10.1097/00004479-200501000-00007. PMID 15682961